CLINICAL TRIAL: NCT00005116
Title: Depression In Juvenile Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: KOVACSM (completed); R01DK025568 (NIH)
Record Dates: First submitted 2000-04-13; First posted 2000-04-14 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Depression; Diabetes Mellitus, Insulin-Dependent
Keywords: depression
MeSH Terms: conditions — Depression; Diabetes Mellitus, Type 1 | interventions — Psychotherapy

INTERVENTIONS:
Behavioral: psychotherapy

SUMMARY:
Depression is one of the most common emotional problems among youths with insulin dependent diabetes mellitus (IDDM). It has been shown that depression in youths with IDDM lasts a while and may have a role in later complications of the medical condition. And yet, there are no psychological interventions appropriate for such youngsters. The purpose of this study is to modify a treatment called ''Contextual Psychotherapy'' (that has been developed for depressed youngsters) in order to address special needs of depressed youths with IDDM, and to ''pilot test'' the treatment. The youngsters to be recruited are those being cared for at the Diabetes Clinic of the Children's Hospital of Pittsburgh. The treatment includes a 3- month phase (16 sessions), followed by a 3-month ''booster'' phase (3 sessions), and two later follow-up evaluations.

ELIGIBILITY:
Inclusion Criteria:

* IDDM duration of less than 10 years
* No major medical disorder other than IDDM
* No psychotropic medications
* Meets psychiatric diagnostic criteria for depression
* Parent and child willing to participate

Exclusion Criteria:

* Does not live withing commuting distance
* Mental retardation

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Maria Kovacs, Principal Investigator — U. Of Pittsburgh School of Medicine
Locations (1):
- WPIC, Pittsburgh, Pennsylvania, United States